CLINICAL TRIAL: NCT00074698
Title: A Phase 1 Study of the Safety, Pharmacokinetics, and Biologic Activity of Escalating Doses of FG-3019 in Subjects With Idiopathic Pulmonary Fibrosis
Brief Title: Safety and Tolerability Study of FG-3019 in Participants With Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FGCL-MC3019-002
Record Dates: First submitted 2003-12-18; First posted 2003-12-22 (Estimated); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic pulmonary fibrosis; IPF; Pulmonary fibrosis; Respiratory disease
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis; Respiration Disorders | interventions — pamrevlumab; Stamulumab

ARMS (3):
- FG-3019 Low Dose (Experimental): Participants will receive a single intravenous (IV) infusion of FG-3019 low dose on Day 0.
  Interventions: Drug: FG-3019
- FG-3019 Medium Dose (Experimental): Participants will receive a single IV infusion of FG-3019 medium dose on Day 0.
  Interventions: Drug: FG-3019
- FG-3019 High Dose (Experimental): Participants will receive a single IV infusion of FG-3019 high dose on Day 0.
  Interventions: Drug: FG-3019

INTERVENTIONS:
Drug: FG-3019 — FG-3019 will be administered per dose and schedule specified in the arm description.
  Other Names: Recombinant human monoclonal antibody

SUMMARY:
The main purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and immunogenicity of FG-3019, a therapeutic antibody designed to block the pro-fibrotic activity of connective tissue growth factor (CTGF). CTGF triggers the production of collagen and fibronectin, which cause scarring and thickening of the lungs. Participants will be assigned sequentially to one of the 3 dose group: Low, medium, and high FG-3019.

ELIGIBILITY:
Key Inclusion Criteria:

* have a diagnosis of idiopathic pulmonary fibrosis (IPF) by clinical features and surgical lung biopsy or according to the American Thoracic Society criteria

Key Exclusion Criteria:

* have a history of significant exposure to organic or inorganic dust or drugs known to cause pulmonary fibrosis
* have interstitial lung disease other than IPF
* have pulmonary fibrosis associated with connective tissue disease
* have other forms of idiopathic interstitial pneumonia, such as desquamative interstitial pneumonia, acute interstitial pneumonia, nonspecific interstitial pneumonia, or cryptogenic organizing pneumonia
* have end-stage IPF (total lung capacity of less than 45% of predicted value)
* are listed for lung transplantation at the time of study enrollment
* have significant heart problems
* are pregnant or lactating (if female)

Other inclusion and exclusion criteria may apply.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2003-12-08 (Actual); Study Completion 2004-05

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Baseline up to 12 months
Area Under the Plasma Concentration Vs Time Curve (AUC) of FG-3019 | Through 30 hours postdose
Number of Participants With Human Anti-human Antibody (HAHA) | Baseline up to 12 months

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - National Jewish Medical and Research Center, Denver, Colorado
  - University of Michigan Health Sciences, Ann Arbor, Michigan
  - Southwestern Medical School, Dallas, Texas
  - University of Washington Medical Center, Seattle, Washington